CLINICAL TRIAL: NCT02272829
Title: Behavioral Consultation for HIV+ Older Adults Prescribed Opioids for Chronic Pain
Acronym: CHOACOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA038203
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Opioid Misuse; Older Adults; HIV
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Active Comparator): Participants in this arm will receive the study intervention (sessions with the BHC and the PCP).
  Interventions: Behavioral: Choacot: Behavioral Intervention for Chronic Opioid Use
- Health Education (Placebo Comparator): Participants in this arm will receive study sessions about various health topics.
  Interventions: Other: Health Education

INTERVENTIONS:
Behavioral: Choacot: Behavioral Intervention for Chronic Opioid Use — This is an intervention for individuals who use opioid medication for chronic pain, and targets the collaboration between the participant and his/her PCP.
  Arms: Active
Other: Health Education
  Arms: Health Education

SUMMARY:
This project will develop a novel collaborative treatment, based on the primary care behavioral consultation model and behavior therapy techniques including motivational interviewing and functional assessment, in which a patient, a Behavioral Health Consultant (BHC) and a HIV primary care provider share a unified plan targeting misuse of prescribed opioid analgesics in older HIV+ adults. The intervention will involve meetings between the BHC and the PCP, the BHC and the participant, and the BHC, PCP and the participant. Opioid misuse will be the primary outcome variable. Quality of the patient-provider relationship, pain, problematic use of other substances, antiretroviral adherence, and psychosocial functioning will be secondary outcomes.

DETAILED DESCRIPTION:
Up to 20% of HIV patients receive prescriptions for chronic opioid therapy (COT) to treat chronic pain. This project will develop a novel collaborative treatment, based on the primary care behavioral consultation model and behavior therapy techniques including motivational interviewing and functional assessment, in which a patient, a Behavioral Health Consultant and a HIV primary care provider share a unified plan targeting misuse of prescribed opioid analgesics in older HIV+ adults. This would be the first theoretically-driven, empirically-tested intervention that specifically attends to the difficult issues around chronic pain and opioid prescription in HIV clinical practice.

This project will develop a collaborative, brief, behavioral consultation intervention targeting misuse of prescribed opioids in older HIV+ adults. The intervention, CHOACOT (Consultation for HIV+ Older Adults on Chronic Opioid Therapy), will consist of:

1. three meetings between the Behavioral Health Specialist (BHS) and the patient
2. two brief consultations between the BHC and the HIV-PCP
3. a joint meeting of the patient, BHC, and HIV-PCP.

To achieve our aims, we will develop CHOACOT beginning with an iterative open trial (n=10). Next, we will conduct a pilot randomized clinical trial (n=30) of CHOACOT versus enhanced Treatment-As-Usual. Opioid misuse will be the primary outcome variable. Quality of the patient-provider relationship, pain, problematic use of other substances, antiretroviral adherence, and psychosocial functioning will be secondary outcomes. The specific aims are:

Aim 1. Develop and refine CHOACOT so that it meets standards of feasibility and acceptability for HIV PCPs, BHCs, and participants;

1a. To develop and field test a CHOACOT BHC manual;

1b. To develop a reliable measure of BHC manual adherence;

1c. To develop and field-test BHC training and supervision procedures. Aim 2. Refine research procedures (e.g., consent and randomization processes, assessment procedures), and establish their feasibility and acceptability to participants while confirming recruitment goal targets.

Misuse of prescribed opioids is the primary outcome. Secondary outcomes are problematic use of substances with a high potential for lethality when used with COT (benzodiazepines, cocaine, alcohol, heroin), ARV adherence, viral load, pain, psychosocial functioning, patient-provider alliance, and treatment satisfaction and acceptability.

This line of work could lead to the incorporation into HIV care of a theoretically-driven and empirically-tested brief intervention for older HIV patients who are prescribed opioids for chronic pain and for whom there is concern about opioid misuse.

ELIGIBILITY:
Inclusion Criteria:

* HIV patients with a physician at the enrollment site;
* Age 50 or older;
* Chronic pain (pain duration for at least six months);
* Daily use of an opioid analgesic, prescribed by an HIV-PCP at the study site, for at least the past 90 days;
* Patients endorse "feeling at risk of losing their pain medication prescription," or that they are "unhappy with how they and their doctors are working together to manage their pain";
* Patient-rated Addictions Behavior Checklist score > 3, as a recommended cut-point indicating opioid misuse.

Exclusion Criteria:

* Current, severe psychiatric symptoms requiring immediate clinical attention;
* Inability to understand English;
* Cognitive impairment severe enough to interfere with ability to actively participate in CHOACOT.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
opioid use | 4 months
  opioid use will be assessed, through self-report measures, monthly over the course of the 4-month study participation period

SECONDARY OUTCOMES:
quality of the patient-provider relationship | 4 months
  quality of the patient-provider relationship will be assessed, through self-report measures, monthly over the course of the 4-month study participation period
pain | 4 months
  pain will be assessed, through self-report measures, monthly over the course of the 4-month study participation period
problematic use of other substances | 4 months
  problematic use of other substances will be assessed, through self-report measures, monthly over the course of the 4-month study participation period
antiretroviral adherence | 4 months
  antiretroviral adherences will be assessed, through self-report measures, monthly over the course of the 4-month study participation period
psychosocial functioning | 4 months
  psychosocial functioning will be assessed, through self-report measures, monthly over the course of the 4-month study participation period

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stein, MD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States